CLINICAL TRIAL: NCT03538665
Title: The DETECT Study - Discovery and Evaluation of Testing for Endometrial and Ovarian Cancer in Tampons: Tampon and Tissue Sampling to Evaluate Markers for Detection of Endometrial and Ovarian Cancer
Brief Title: The DETECT Study: Discovery and Evaluation of Testing for Endometrial and Ovarian Cancer in Tampons
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rebecca Arend, Associate Professor, University of Alabama at Birmingham
Other Study IDs: 999918106; Z01CP010124-21 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-05-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer; Endometrial Cancer Precursors; Ovarian Cancer; Complex Atypical Endometrial Hyperplasia
Keywords: Endometrial Cancer; Somatic Mutations; Early Detection; Tampon Sampling; Tissue Discovery; Natural History; Ovarian Cancer; Screening Tool
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Women undergoing clinically-indicated hysterectomy +/- bilateral salpingo-oophorectomy for endometrial or ovarian cancer or precursors
- Controls: Women undergoing clinically-indicated hysterectomy for benign conditions

SUMMARY:
BACKGROUND:

Endometrial cancer is a common and deadly cancer for women. It is getting more common and deadly because risk factors like age and obesity are increasing. Also, this cancer is becoming more common and deadly for black women than white women. Researchers want to find better ways to take samples and test them for this cancer. They want to study this for a racially diverse population. One way to take samples might be from a tampon. If identified early, endometrial cancer can be highly curable; however, the earliest stages may be asymptomatic, and clinical symptoms are often missed. Combining sensitive molecular testing approaches with non-invasive sampling techniques may to lead to the development of novel endometrial cancer early detection approaches with the potential to overcome disparities in access to care and time to diagnosis and treatment.

In contrast to endometrial cancer, ovarian cancer is typically detected at advanced stages with poor survival since symptoms manifest only late in the disease process and are very unspecific. Racial disparities in ovarian cancer incidence and mortality are also much less pronounced. Racial disparities can manifest particularly when screening, symptom appraisal and early detection, and effective treatment interventions have important roles in determining outcomes of cancers.

OBJECTIVES:

The purpose of this study is to see if it is possible and acceptable for individuals to have an endometrial or ovarian sample collected by using a tampon placed in the vagina. The investigators will look at DNA in these samples. DNA is the genetic information participants inherited from their parents. The investigators want to see whether the investigators can find changes in DNA and proteins related to endometrial or ovarian cancer from tampon samples. Tests on the samples from tampons will help to understand endometrial and ovarian cancer. The samples collected during this study will be used for research related to both endometrial and ovarian cancer and non-cancer conditions.

ELIGIBILITY:

Women at least ≥18 years undergoing clinically-indicated hysterectomy and/or bilateral salpingo-oophorectomy for endometrial or ovarian cancer, cancer precursors, or benign conditions.

DESIGN:

1. Participants will put a tampon in their vagina at least 30 minutes before their surgery.
2. Participants will take a short survey.
3. The tampon will be collected during the surgery.
4. A small piece of tissue will be collected from the uterus +/- ovary that is removed in surgery.
5. Participants will give a blood sample.
6. Before or after surgery, participants will answer questions. These will be about their medical history and basic data such as age and race.
7. Researchers will follow participants medical records for up to 5 years after the study. Additional blood may be taken from patient if patient agrees.
8. Researchers will study the samples and tampons. They will compare how well cancer and other markers are detected between the samples.

DETAILED DESCRIPTION:
BACKGROUND:

Endometrial cancer is the most common and second deadliest gynecological cancer in women in the United States, with over 65,000 new cases and 12,000 deaths expected to occur in 2022. Unlike most cancers, endometrial cancer incidence and mortality are increasing, due primarily to rising rates of aggressive subtypes of endometrial cancer (non-endometroid tumors, i.e., serous or clear cell histology), which are more common in Black or African American (henceforth referred to as "Black") women. In addition to being more clinically aggressive, these non-endometrioid tumors are thought to have different risk factor profiles, precursor lesions, and molecular features than the more common and less aggressive endometrioid subtypes.

The same morphologic subtypes (serous and endometrioid) with similar molecular profiles are also found in ovarian cancers, which share many risk factors with endometrial cancers.

Racial disparities in endometrial cancer incidence and mortality have been reported, with Black women experiencing more rapid increases in incidence, as well as a higher burden of endometrial cancer mortality compared to other racial/ethnic groups. The underlying basis for these disparities is likely multifactorial, involving biological differences, as well as clinical factors related to access to care, delayed diagnosis, and differences in treatment and surgical management.

If identified early, endometrial cancer can be highly curable; however, the earliest stages may be asymptomatic, and clinical symptoms are often missed. Combining sensitive molecular testing approaches with non-invasive sampling techniques may to lead to the development of novel endometrial cancer early detection approaches with the potential to overcome disparities in access to care and time to diagnosis and treatment.

In contrast to endometrial cancer, ovarian cancer is typically detected at advanced stages with poor survival since symptoms manifest only late in the disease process and are very unspecific. Racial disparities in ovarian cancer incidence and mortality are also much less pronounced. Racial disparities can manifest particularly when screening, symptom appraisal and early detection, and effective treatment interventions have important roles in determining outcomes of cancers. Contrasting ovarian and endometrial cancers, which have similar risk factors and biologic underpinnings, but very different clinical courses, can further help to elucidate the role of behavioral and healthcare system-related causes of endometrial cancer disparities.

The investigators and others have recently shown that lower genital tract sampling approaches such as vaginal tampons, offer an acceptable and feasible method for identifying molecular markers with high sensitivity and specificity for endometrial and ovarian cancers. Importantly, these proof-of-principle studies have been conducted in predominantly non-Hispanic white (white) populations, and studies of molecular markers for endometrial and ovarian cancer, including those involving vaginal tampons, are lacking in black women.

OBJECTIVES:

The primary objectives of this study are to Aim 1) Characterize racial differences in risk factor associations with endometrial and ovarian cancers by histologic subtype; Aim 2) Assess associations of care delays related to symptom appraisal with endometrial cancer diagnosis and whether delays are associated with tumor characteristics; Aim 3) Evaluate determinants of acceptability and feasibility of vaginal tampon sampling; 4) Evaluate the performance of molecular biomarkers for endometrial cancer detection in paired tampon-collected and tissue specimens, overall and by race and histologic subtype; 5)Evaluate clinical, molecular, and epidemiological factors associated with endometrial cancer recurrence and survival overall and by race.

The secondary objective of this study are to: 1) Compare findings in ovarian cancer cases and controls to findings in endometrial cancer cases and controls as described in primary aims 1-5. For each specific aim above, ovarian cancer will represent an important comparison to (1) understand novel risk factor and biological associations by comparing histologic subtypes across cancer sites, (2+3) to better understand the role of behavioral and healthcare system-related causes of endometrial cancer disparities, (4) to evaluate biomarkers for gynecological cancer detection, and (5) to study factors associated with prognosis and outcomes; 2) Support discovery and validation efforts of liquid biopsy markers and artificial intelligence approaches for prognostic applications.

The goal of this study is to evaluate the acceptability, feasibility, and clinical performance of vaginal tampon sampling for molecular testing of endometrial cancer early detection biomarkers in a racially diverse clinical population.

ELIGIBILITY:

Eligible participants will include people with a uterus (hereafter referred to as "women") aged ≥18 years undergoing clinically-indicated hysterectomy and/or bilateral salpingo-oophorectomy for endometrial or ovarian cancer, cancer precursors, or benign conditions at the University of Alabama's Division of Gynecologic Oncology and Department of Gynecology.

DESIGN:

This is a case-control study with prospective follow-up of the electronic health record for up to 5 years. Cases will be defined as women with histologically-confirmed endometrial or ovarian cancer or cancer precursors diagnosed at hysterectomy/oophorectomy. Controls will have no histologic evidence of endometrial or ovarian cancer or cancer precursors diagnosed at hysterectomy/oophorectomy.

The primary endpoints of this study will be: 1) Associations of clinical and epidemiologic factors with odds of endometrial and ovarian cancer by race and subtype; 2) Associations of factors related to symptom appraisal and care delay with tumor characteristics, overall and by race; 3) The acceptability and feasibility of vaginal tampon sampling, assessed by evaluating 10 items from a brief survey regarding tampon sampling and the DNA yield from the vaginal tampon, respectively; 4) The prevalence, sensitivity, and specificity of endometrial and ovarian cancer molecular biomarkers in tampon and tissue samples in cases and controls; 5) Associations of clinical, molecular, and epidemiologic predictors of endometrial and ovarian cancer recurrence and survival.

ELIGIBILITY:
INCLUSION CRITERIA:

* Individuals born with female sex organs (uterus, ovaries, including cis-gender female and transmasculine individuals, hereafter referred to as "women") scheduled for hysterectomy or bilateral salpingo-oopherectomy at the University of Alabama Birmingham's Division of Gynecologic Oncology or Department of Gynecology
* Age >18 years. We have chosen this age range to include both peri- and postmenopausal women, who are at greatest risk for endometrial cancer.
* Ability of study participant to understand and the willingness to sign a written informed consent document. Women who do not meet this criterion include potential participants who do not speak English or Spanish, or have physical, mental, or emotional problems that prevent them from comprehending the nature of the study. If the potential participant has trouble reading the document, the designated study staff person may read the document to the patient, to include the basic elements of the informed consent document, per 45 CFR §46.116 (a).

EXCLUSION CRITERIA:

* Women who are pregnant are excluded from gynecologic surgery and are therefore not eligible to participate.
* Individuals who were not born with female sex organs at birth (i.e., cis-gender males and transfeminine individuals) are not eligible for this study as they are not at risk for developing endometrial and ovarian cancer.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals >18 years of age born with female sex organs (uterus, ovaries, including cis-gender female and transmasculine individuals, hereafter referred to as "women") scheduled for hysterectomy or bilateral salpingo-oopherectomy at the University of Alabama Birmingham's Division of Gynecologic Oncology or Department of Gynecology.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Endometrial Cancer | Enrollment or at time of surgery
  Women with histologically confirmed diagnosis of endometrial or ovarian cancer
Endometrial cancer precursors | Enrollment or at time of surgery
  Women with histologically confirmed diagnosis of precursors (e.g., atypical hyperplasia)
Non-malignant uterus | Enrollment or at time of surgery
  Women with fibroids, polyps, endometrial hyperplasia without atypia, adenomyosis, normal endometrium, or other benign conditions determined by histology and/or clinical imaging.

SECONDARY OUTCOMES:
Acceptability of tampon sampling | Prior to surgery
  Women will be given a 10 question survey to assess acceptability of tampon sampling
Feasibility of tampon sampling | During and immediately after surgery
  The feasibility of tampon sampling will be determined by successful tampon insertion according to protocol prior to surgery and sufficient DNA yield (e.g., 1-2 microgram) from the tampon sample.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Arend, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Bakkum-Gamez JN, Wentzensen N, Maurer MJ, Hawthorne KM, Voss JS, Kroneman TN, Famuyide AO, Clayton AC, Halling KC, Kerr SE, Cliby WA, Dowdy SC, Kipp BR, Mariani A, Oberg AL, Podratz KC, Shridhar V, Sherman ME. Detection of endometrial cancer via molecular analysis of DNA collected with vaginal tampons. Gynecol Oncol. 2015 Apr;137(1):14-22. doi: 10.1016/j.ygyno.2015.01.552. Epub 2015 Feb 10. PMID 25677060
- [Background] Erickson BK, Kinde I, Dobbin ZC, Wang Y, Martin JY, Alvarez RD, Conner MG, Huh WK, Roden RBS, Kinzler KW, Papadopoulos N, Vogelstein B, Diaz LA Jr, Landen CN Jr. Detection of somatic TP53 mutations in tampons of patients with high-grade serous ovarian cancer. Obstet Gynecol. 2014 Nov;124(5):881-885. doi: 10.1097/AOG.0000000000000484. PMID 25437714
- [Background] Nair N, Camacho-Vanegas O, Rykunov D, Dashkoff M, Camacho SC, Schumacher CA, Irish JC, Harkins TT, Freeman E, Garcia I, Pereira E, Kendall S, Belfer R, Kalir T, Sebra R, Reva B, Dottino P, Martignetti JA. Genomic Analysis of Uterine Lavage Fluid Detects Early Endometrial Cancers and Reveals a Prevalent Landscape of Driver Mutations in Women without Histopathologic Evidence of Cancer: A Prospective Cross-Sectional Study. PLoS Med. 2016 Dec 27;13(12):e1002206. doi: 10.1371/journal.pmed.1002206. eCollection 2016 Dec. PMID 28027320